CLINICAL TRIAL: NCT04072640
Title: The Effect and Safety of Three Initial Introduction Treatments on HIV-infected Patients With Cryptococcal Meningitis: A Multi-center, Random and Prospective Study
Brief Title: Three Induction Treatments on Cryptococcal Meningitis
Acronym: TITOC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Wenzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-014-1
Record Dates: First submitted 2019-06-09; First posted 2019-08-28 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Cryptococcal Meningitis; HIV/AIDS
Keywords: Voriconazole;amphotericin ;cryptococcal meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal; Acquired Immunodeficiency Syndrome | interventions — Voriconazole; amphotericin B, deoxycholate drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- voriconazole treatment (Experimental): induction treatment with Voriconazole 200mg bid (IV) + 5FC (100mg/kg/d) for 14 days, consolidation treatment wiht fluconazole 400mg/d for two months, then maintenance treatment with fluconazole 200mg/d
  Interventions: Drug: Voriconazole 200mg
- amphotericin treatment (0.7-1.0mg/kg/d) (Active Comparator): Induction treatment with amphotericin B 0.7-1.0mg/kg/d + 5FC (100mg/kg/d) for 14 days,consolidation treatment wiht fluconazole 400mg/d for two months, then maintenance treatment with fluconazole 200mg/d
  Interventions: Drug: Amphotericin B-deoxycholate (0.7-1.0mg/kg/d)
- amphotericin B treatment (0.4-0.5mg/kg/d) (Experimental): Induction treatment with amphotericin B 0.4-0.5mg/kg/d + 5FC (100mg/kg/d) for 28 days, consolidation treatment with fluconazole 400mg/d for two months, then maintenance treatment with fluconazole 200mg/d
  Interventions: Drug: amphotericin B deoxycholate (0.4-0.5mg/kg/d)

INTERVENTIONS:
Drug: Voriconazole 200mg — Induction treatment with voriconazole( 400mg/d)+5FC (100mg/kg/d) for 14 days;
  Other Names: Voriconazole for Cryptococcus
  Arms: voriconazole treatment
Drug: amphotericin B deoxycholate (0.4-0.5mg/kg/d) — Induction treatment with 0.4-0.5mg/kg/d of Amphotericin B-deoxycholate +5FC(100mg/kg/d) for 28 days
  Other Names: low dose and long course of Amphotericin B-deoxycholate
  Arms: amphotericin B treatment (0.4-0.5mg/kg/d)
Drug: Amphotericin B-deoxycholate (0.7-1.0mg/kg/d) — Induction treatment with 0.7-1.0mg/kg/d of Amphotericin B-deoxycholate +5FC(100mg/kg/d) for 14 days
  Other Names: standard Amphotericin B-deoxycholate for Cryptococcus
  Arms: amphotericin treatment (0.7-1.0mg/kg/d)

SUMMARY:
Three induction treatment strategies [ voriconazole +5FC vs. amphotericin deoxycholate (0.4-0.5 mg/kg/d)+5FC vs. amphotericin deoxycholate (0.7-1.0 mg/kg/d)+5FC ] for HIV-infected patients with cryptococcal meningitis were compared.

DETAILED DESCRIPTION:
HIV-associated cryptococcal meningitis were randomly allocated into three induction treatment as follow: 1) 14 days of voriconazole 200mg bid +5FC, 2) 28 days of amphotericin deoxycholate (0.4-0.5 mg/kg/d) +5FC ; 3）14 days of deoxycholate (0.7-1 mg/kg/d) +5FC). After induction treatment were finished, all groups switched into fluconazole(400mg/d) for two-month consolidation treatment. 14-day early fungicidal rate, 90-day mortality, side effects , and tolerances were compared between three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of HIV infection;
2. newly diagnosed Cryptococcal Meningitis by positive India ink staining or culture result, or both in cerebrospinal fluid (CSF);
3. Anti-viral treatment naïve patients
4. anti-fungal treatment naïve patients

Exclusion Criteria:

1. hepatitis virus co-infection;
2. liver cirrhosis;
3. congestive heart failure;
4. chronic renal disorders;
5. chronic obstructive pulmonary disease (COPD);
6. Tuberculosis co-infection;
7. malignances
8. severe mental and neurological diseases
9. Women during pregnancy and lactation
10. intraveneous drug user (IDU)
11. patients with follow abnormal test results:hemoglobin < 6 g/dl, white blood cell count < 2000 / μl, neutrophil count < 1000 / μl, platelet count < 75000 / μl, blood amylase > 3 times normal level Upper limit, serum creatinine > 1.5 times normal upper limit, aspartate aminotransferase / alanine aminotransferase / alkaline phosphatase > 3 times normal upper limit, total bilirubin > 2 times normal upper limit
12. patients who are unwilling to anticipate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
90-day Cryptococcal Meningitis (CM) related mortality | 90 days
  analysis of 90-day CM-related mortality of patients in three induction treatments

SECONDARY OUTCOMES:
Early fungicidal rate in Cerebrospinal fluid (CSF) | 2 weeks
  Comparison of 2-week CSF early fungicidal activity in three induction treatments
creatinine elevation | 0-90 days
  TO observe the numbers of patients whose creatinine > 110 mmol/L during antifungal therapy
Hypokalemia | 0-90 days
  To observe the rate of hypokalemia in three groups during antifungal therapy
anemia | 0-90 days
  Comparison of the numbers of patients with hemoglobin <120g/L for male or <110g/L for female.

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Xu, PH.D, Principal Investigator — Zhejiang University
Locations (1):
- Lijun Xu, Zhenjiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
12 months after study finished
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months
Access Criteria: Qualified researchers may submit a request containing the research objectives, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s).